CLINICAL TRIAL: NCT04725916
Title: Studying How Outpatient Water affEcts Risks With Drains (SHOWER Study)
Acronym: SHOWER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sean Devitt (Other)
Responsible Party: Sponsor-Investigator, Sean Devitt, Sponsor-Investigator, Geisinger Clinic
Organization: Geisinger Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0970
Record Dates: First submitted 2021-01-20; First posted 2021-01-27 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Wound Infection; Postoperative Complications; Surgical Site Infection; Drain Site Complication
Keywords: Panniculectomy; Breast reduction surgery; Postoperative showering; Surgical drain; Fleur-de-lis panniculectomy; Massive weight loss surgery
MeSH Terms: conditions — Surgical Wound Infection; Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Arm 1 (Active Comparator): Subjects assigned to Arm 1 will be instructed to shower daily beginning on post-operative Day 2 and maintain this daily schedule until the subject's 3-month standard of care clinic follow-up visit. They will receive specific instructions on caring for the incision site and drains until they are removed.
  Interventions: Other: Showering
- Study Arm 2 (Active Comparator): Subjects assigned to Arm 2 will be instructed not to shower post-operatively until their surgical drains are removed. They will receive specific instructions on bathing and caring for the incision sites and drains.
  Interventions: Other: Restriction of Showering

INTERVENTIONS:
Other: Showering — Patients will be instructed to shower after surgery with drains in place
  Arms: Study Arm 1
Other: Restriction of Showering — Patients will be restricted from showering post operatively if they have drains in place
  Arms: Study Arm 2

SUMMARY:
This is a prospective randomized, controlled, unblinded, interventional feasibility study to evaluate if showering with post operative drains in place leads to an increase in complications. The patients included in the study will be those undergoing breast reductions and panniculectomies at Geisinger Medical Center. The patients will be randomized post operatively into one of two groups: 1) patients instructed to shower with drains in place, and 2) patients instructed not to shower while they have drains in place.

DETAILED DESCRIPTION:
This is a prospective randomized, controlled, unblinded interventional feasibility trial evaluating the post-operative outcomes of surgical patients undergoing breast reduction or panniculectomy procedures. Approximately 100 eligible subjects will undergo their surgical procedure according to standard clinical guidelines. Unless clinically contraindicated, study surgeons will maintain consistent use of 10 Flat drains for all study participants to prevent any sampling bias.

Immediately after surgery is completed, the study investigator will randomize the subject into one of the 2 study arms. The randomization scheme will control for procedure type.

The study will not be blinded. The randomization assignment will be communicated to the care team and documented in the subject's electronic medical record to ensure that appropriate post-operative instruction is provided to the subject. Subjects will be notified of their study arm assignment at the time they receive their post-operative discharge instruction.

Subjects in both arms will complete a questionnaire related to quality of life post-operatively, as well as daily bathing specifics.

The following statistical methods will be used for the aims:

Aim 1: Collect and describe information related to outcome measures in addition to study data including number eligible, response rates, adherence/compliance rates.

Descriptive statistics will be provided for all study enrollment data, compliance information as well as data collected throughout the study including outcome measures and responses from the satisfaction survey.

Aim 2: To compare the surgical site complication rate of post-operative patients with drains who shower versus those who do not shower.

Complication rates between the two study arms will be compared using chi-squared tests, although these comparisons will not be conclusive since the study isn't powered to assess equivalence.

Aim 3: To compare patient post-operative satisfaction for those who shower versus those who do not shower.

Patient post-operative satisfaction between the two study arms will be compared using chi-squared tests, although these comparisons will not be conclusive since the study isn't powered to assess differences.

ELIGIBILITY:
Inclusion Criteria:

* Patients having one of the following procedures at Geisinger Medical Center in which drains are placed

  * Breast reduction
  * Lower panniculectomy
  * Fleur-de-lis panniculectomy
* ≥18 years of age
* Able and willing to provide consent

Exclusion Criteria:

* Patients on antibiotics at the time of surgery
* Patients sent home on antibiotics after surgery
* Patients who work in healthcare with direct patient contact
* Patients having a panniculectomy to be eligible for a kidney transplant
* Patients having a ventral hernia repair at the time of the panniculectomy
* Patients admitted to the hospital for >1 night

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Drain site cellulitis | 12 weeks
  At each post operative appointment, the patient's drain sites will be examined for signs of cellulitis including tenderness to palpation and blanching erythema. The decision will be based on clinical exam by the physicians assistant, confirmed with the attending physician, and photos will be taken for documentation.
Incisional cellulitis | 12 weeks
  At each post operative appointment, the patient's incision will be examined for signs of cellulitis including tenderness to palpation and blanching erythema. The decision will be based on clinical exam by the physicians assistant, confirmed with the attending physician, and photos will be taken for documentation.
Seroma formation | 12 weeks
  At each post operative visit, the patient will be examined to rule out the presence of wound seroma. Any seroma requiring needle aspiration with removal of fluid will be documented as a positive seroma.
Abscess formation | 12 weeks
  The patient will be examined at each post operative visit. Any collection of bacteria (abscess) that requires bedside drainage will be recorded as an abscess.
Wound dehiscence | 12 weeks
  Development of wound dehiscence during follow-up period
Patient Satisfaction | 12 weeks
  Measurement of patient satisfaction of post-operative ability to shower based on administration of a satisfaction survey

CONTACTS AND LOCATIONS:
Overall Officials: Sean Devitt, MD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No